CLINICAL TRIAL: NCT06791564
Title: Minimally Invasive Active Release of Septa Bands for Cellulite and Connective Tissue Release for Fibrosis Treatment in Body Contouring Surgery
Acronym: AVE001
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Total Definer Research Group (Other)
Responsible Party: Principal Investigator, Alfredo Hoyos, MD, Plastic Surgeon | Total Definer, Total Definer Research Group
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aveli
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Liposuction; Cellulite; Cellulite Reduction; Fibrosis; Skin
Keywords: Aveli; Body contouring; Liposuction; Liposculpture; Cellulite reduction; Fibrosis Reduction; Fibrotic tissue
MeSH Terms: conditions — Cellulite; Fibrosis

STUDY DESIGN:
Intervention Model Description: All the participants are categorized into the 3 different intervention groups based on the individual pre-procedure physical exam by the plastic surgeon. Once in the study group, the patient receives the intervention corresponding to this arm of the study.
Masking Description: No masking was feasible for this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cellulite group (CG) (Experimental): Patients with any degree of clinically evident cellulite undergoing HDL + AVÉLI treatment for Cellulite.
  Interventions: Device: AVELI
- Fibrosis Group (FG) (Experimental): Patients with any degree of fibrosis undergoing non-primary HDL + AVÉLI release of fibrotic tissue.
  Interventions: Device: AVELI
- Fibrosis and Cellulite Group (FCG) (Experimental): Patients with any degree of clinically evident cellulite AND fibrosis undergoing non-primary HDL + AVÉLI treatment for both.
  Interventions: Device: AVELI

INTERVENTIONS:
Device: AVELI — Minimally invasive method for selectively identifying and manually releasing specific septa responsible for causing cellulite depressions.

SUMMARY:
This prospective study aims to evaluate the safety and effectiveness of AVELI for reducing cellulite and fibrotic tissue in patients undergoing High-Definition Liposculpture, exploring if AVELI improves the aesthetic outcomes, and reduced the clinically evident cellulite and/or fibrosis.

The main questions this study seeks to answer are:

* Does AVELI safely reduce cellulite and fibrotic tissue without causing serious adverse events?
* How effective is AVELI in improving patient-reported outcomes and aesthetic appearance?

Through this study, the study team aims to evaluate the safety and effectiveness of AVELI.

The study procedures include:

* Baseline data collection of sociodemographic variables. Data collection of surgical variables, adverse events, and satisfaction scores.
* All patients will undergo the standardized High-Definition Liposculpture technique, with AVELI applied to all identified cellulite and/or fibrosis release.
* Photographic and 3D imaging preoperatively and at follow-ups (1, 3, 6, and 9 months).

DETAILED DESCRIPTION:
Study design: Interventional prospective cohort study, non-randomized, non-controlled, no masking.

Ethical Considerations:

* IRB Approval: The study will adhere to the Declaration of Helsinki principles and will be approved by an Institutional Review Board (IRB).
* Informed Consent: Participants will be provided comprehensive information about study procedures, risks, and benefits, and written consent will be obtained.
* Data Confidentiality: All participant data will be anonymized and securely stored.

Eligible patients will be approached, the study aims, objectives, procedures, and voluntary participation will be explained. In case patient consent to participate, a written informed consent will be signed. The patients will be comprehensively evaluated by the plastic surgeon, and assigned to a group based on their individual physical evaluation findings: Cellulite Group, Fibrosis Group, Fibrosis and Cellulite Group.

Study Locations:

* Dhara Clinic (Bogota, Colombia)
* Miami Aesthetic Center (Miami, FL - USA)

Data Collection:

* Demographic, Clinical, and surgical variables are going to be collected in an Excel-based password protected database.
* Other procedure related variables are also going to be collected in the same database, including pain assessment in the immediate postoperative, hemoglobin and hematocrit levels, time to discharge, and complications & management.
* 3D photographic analysis will be employed to analyze preoperative, and postoperative images at 1, 3, 6 and 9 months post procedure. Then the changes will be objectively compared using Quantificare Photographical Software, through the different timepoints to evaluate the objective contour defects and postoperative improvement changes.
* Satisfaction Scores: Global Aesthetic Improvement Scale (GAIS) evaluated at least 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing HDL between 18 and 60 years old.
* Non-gender specific.
* American Association of Anesthesiologist Risk Assessment (ASA) ≤ 2.
* Body Mass Index (BMI) ≥20 and ≤ 32 kg/m2.
* Patients with any degree of clinically evident cellulite in any body area.
* Patients with prior liposuction procedures with any degree of fibrosis in any body area.
* Patients undergoing additional procedures such as, but not limited to: Rhinoplasty, Mammaplasty, Mastopexy, mini tummy tuck, full tummy tuck, brachioplasty, thighplasty, fat grafting. The procedure could not be related to the treatment of fibrosis or cellulite.

Exclusion Criteria:

* Patients requiring SQ fat grafting for the amendment of any contour irregularity.
* Patients requiring other devices/drugs for skin contraction and/or cellulite treatment for the next 6 months (RF, US, Enzymes, etc.).
* Patients undergoing Face Lift procedures.
* Patients with any history of abnormal scarring and/or hypertrophic scars and or keloids.
* Patients with Caprini score ≥ 8.
* Patients with past medical history of connective tissue disease with active disease and/or recent relapse.
* Patients with past medical history thromboembolic disease or any other condition with an increased risk of coagulopathy (i.e., SLE, RA, APS).
* Patients using aspirin or any anticoagulant within 14 days and 5 days prior to surgery, respectively.
* Patients with a PMH of epilepsy or any epileptic syndrome and or vascular disease.
* Patients with any chronic disease non-compliant with treatment or non-adequately controlled.
* Positive pregnancy test or planning on getting pregnant in the next 6 months.
* Patients with fever or any other symptoms/signs of infection.
* Active smokers or chronic smokers with recent quit (≤ 4-8 weeks).
* Patients with prothrombin time (PT) and/or activated partial thromboplastin time (aPTT) >1.5 times baseline.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events Incidence | 30 days
  Incidence of intervention-related serious adverse events (SAE). SAE were defined as any adverse events that met one or more of the following criteria: required hospital care, required additional medical intervention or treatment, produced any disability, were classified as life-threatening, or resulted in the death of the patient.
Patient Satisfaction Scores | 6 months
  Patient-reported satisfaction scores measured using Global Aesthetic Improvement Scale (GAIS) for the reduction of cellulite and/or fibrosis.
  The GAIS is a standardized scale used primarily in cosmetic and dermatological treatments to assess the overall aesthetic improvement of a patient after a procedure. It consist of three questions:
  * how do you feel about your appearance after surgery? Possible answers: Very much improved, much improved, slightly improved, no change.
  * Are you satisfied with the surgery? Very satisfied, satisfied, not satisfied.
  * Would you recommend the surgical procedure? Possible answers: Yes, perhaps, no.
Photographic aesthetic outcomes analysis | One month, three months, six months, and nine months
  Through 3D camera photos and photographic software, an analysis will objectively calculate the differences between preoperative contour defects (fibrosis and/or cellulite) and postoperative improvement.

CONTACTS AND LOCATIONS:
Locations (2):
- Miami Aesthetic, Miami, Florida, United States
- Dhara Clinic, Bogotá, DC, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Depending upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: After results publication (manuscript)
Access Criteria: Request to the main author

REFERENCES:
- [Background] Stevens WG, Green JB, Layt C, Kaminer MS, Harrington J, Fan L, Wall HC, Fabi S, Magnusson MR. Multicenter Pivotal Study Demonstrates Safety and Efficacy of a New Cellulite Procedure: Final Results at 12 Months. Aesthet Surg J. 2023 Mar 15;43(4):455-466. doi: 10.1093/asj/sjac291. PMID 36351188
- [Background] Stevens WG, Kaminer MS, Fabi SG, Fan L. Study of a New Controlled Focal Septa Release Cellulite Reduction Method. Aesthet Surg J. 2022 Aug 1;42(8):937-945. doi: 10.1093/asj/sjac010. PMID 35089992
- [Background] Danilla S, Babaitis RA, Jara RP, Quispe DA, Andrades PR, Erazo CA, Albornoz CR, Sepulveda SL. High-Definition Liposculpture: What are the Complications and How to Manage Them? Aesthetic Plast Surg. 2020 Apr;44(2):411-418. doi: 10.1007/s00266-019-01475-6. Epub 2019 Aug 20. PMID 31432229
- [Background] Bass LS, Kaminer MS. Insights Into the Pathophysiology of Cellulite: A Review. Dermatol Surg. 2020 Oct;46 Suppl 1(1):S77-S85. doi: 10.1097/DSS.0000000000002388. PMID 32976174
- [Background] Friedmann DP, Vick GL, Mishra V. Cellulite: a review with a focus on subcision. Clin Cosmet Investig Dermatol. 2017 Jan 7;10:17-23. doi: 10.2147/CCID.S95830. eCollection 2017. PMID 28123311
- [Background] Gabriel A, Chan V, Caldarella M, Wayne T, O'Rorke E. Cellulite: Current Understanding and Treatment. Aesthet Surg J Open Forum. 2023 Jun 21;5:ojad050. doi: 10.1093/asjof/ojad050. eCollection 2023. PMID 37424836
- [Background] Ferry AM, Chamata E, Dibbs RP, Rappaport NH. Avoidance and Correction of Deformities in Body Contouring. Semin Plast Surg. 2021 May;35(2):110-118. doi: 10.1055/s-0041-1727207. Epub 2021 Jun 8. PMID 34121946